CLINICAL TRIAL: NCT02323269
Title: A Multicenter, Open-Label, 12-Month Observational Study Evaluating the Clinical Effectiveness and Impact on Patient-Reported Outcomes of Oral Tecfidera™ (Dimethyl Fumarate) Delayed-Release Capsules in Patients With Relapsing-Remitting Multiple Sclerosis, Who Are Either Treatment-Naïve or Switching From an Interferon or Glatiramer Acetate After Suboptimal Response (ImPROve)
Brief Title: Effectiveness of DMF (Dimethyl Fumarate) and Its Impact on PROs (Patient Reported Outcomes) in Treatment-Naive or Suboptimal IFN (Interferon) or GA (Glatiramer Acetate) Responders With RRMS (ImPROve)
Acronym: IMPROVE
Status: Terminated | Type: Observational
Why Stopped: 109MS415 ImPROve study was terminated due to patient enrollment challenges and feasibility . The decision was not a result of safety concerns.
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: 109MS415; CAN-BGT-14-10614 (Other: Sponsor)
Record Dates: First submitted 2014-12-18; First posted 2014-12-23 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-04

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting; Relapsing-Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Dimethyl Fumarate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Treatment naive to dimethyl fumarate: Participants who are prescribed dimethyl fumarate as their initial therapy will receive 120 mg tablet administered orally twice a day for 7 days, then switch to maintenance dose of 240 mg tablet twice daily.
  Interventions: Drug: dimethyl fumarate
- Switch to dimethyl fumarate: Participants who are prescribed dimethyl fumarate after suboptimal response to IFN or GA will receive 120 mg tablet administered orally twice a day for 7 days, then switch to maintenance dose of 240 mg tablet twice daily.
  Interventions: Drug: dimethyl fumarate

INTERVENTIONS:
Drug: dimethyl fumarate — administered according to the local product label (i.e., Canadian Product Monograph).
  Other Names: DMF; BG00012; Tecfidera

SUMMARY:
The primary objective of the study is to estimate the annualized relapse rate (ARR) over a 12-month period in patients with Relapsing-Remitting Multiple Sclerosis (RRMS) who are treated with dimethyl fumarate (DMF) as their initial therapy (treatment-naïve), or switching from interferon (IFN) or glatiramer acetate (GA) (after suboptimal response defined as suboptimal efficacy, intolerance, or poor adherence to IFN or GA), as determined by the Prescribing Physician. The secondary objectives of this study in this study population are: To assess the impact of DMF over a 12 month period on patient reported outcomes (PROs) and health economic related outcomes; and to evaluate additional clinical outcomes at Month 12.

ELIGIBILITY:
Key Inclusion Criteria:

* Have access to the internet and are able to complete online assessments on a computer.
* Have relapsing-remitting MS and satisfy the approved therapeutic indication for DMF per the Canadian Product Monograph.
* Are either treatment-naïve or being treated for RRMS with IFN or GA but, per the Prescribing Physician, have a suboptimal response (e.g., suboptimal efficacy, intolerance, or poor adherence) to IFN or GA or have stopped treatment with IFN or GA for RRMS as a result of suboptimal response within 30-60 days of enrollment.

Key Exclusion Criteria:

* Have major comorbid conditions that would preclude their participation in the study as determined by the Prescribing Physician.
* Have a history of malignancy. (Patients with basal cell carcinoma that has been completely excised prior to study entry remain eligible.)
* Are receiving disease modifying therapies other than IFN or GA or have initiated treatment with a new disease modifying therapy since discontinuation of IFN or GA.

NOTE: Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be conducted in male and female patients with relapsing-remitting MS who satisfy the therapeutic indication for DMF per the Canadian Product Monograph, and who are either treatment-naïve or responding suboptimally to MS platform therapies (e.g., IFN or GA), as determined by the Prescribing Physician.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2015-05; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Annualized Relapse Rate (ARR) at month 12 | Month 12
  Relapses are defined as new or recurrent neurologic symptoms not associated with fever, lasting at least 24 hours.

SECONDARY OUTCOMES:
Change from baseline to Month 12 in the 14-item Treatment Satisfaction Questionnaire for Medication (TSQM-14) score | Baseline and month 12
  TSQM-14 is an instrument to assess patient's satisfaction with medication, providing scores on four scales: Side effects, effectiveness, convenience and global satisfaction.
Change from baseline to Month 12 in the Short-Form 36 (SF-36) scores | Baseline and month 12
  SF-36 is a self-administered, generic health status questionnaire consisting of 36 questions that measure 8 health concepts: physical functioning, role limitations due to physical problems, bodily pain, general health perception, vitality, social functioning, role limitations due to emotional problems and mental health.
Change from baseline to Month 12 in the Modified Fatigue Impact Scale (MFIS-5) scores | Baseline and month 12
  MFIS-5 a modified form of the Fatigue Impact Scale that consists of five questions that assess the impact of fatigue on physical, cognitive, and psychosocial functioning, with five response levels ranging from 0 ("Never") to 4 ("Almost always"). Total scores range from 0 to 20, with higher scores representing a greater impact of fatigue.
Change from baseline to Month 12 in the Beck Depression Inventory (BDI-7) scores | Baseline and month 12
  BDI-7 is is a self-report inventory for measuring the severity of depression on a 7-item scale.
Change from baseline to Month 12 in the Work Productivity and Impairment Questionnaire: Multiple Sclerosis (WPAI-MS) scores | Baseline and month 12
  WPAI-MS is a patient-reported quantitative assessment of the amount of absenteeism, presenteeism and daily activity impairment attributable to Multiple Sclerosis
Change from baseline to Month 12 in the Morisky 8-item Medication Adherence Scale (MMAS-8) scores | Baseline and month 12
  MMAS-8 is a self-reporting tool to facilitate the identification of barriers to and behaviors associated with adherence to chronic medications. Scores on the MMAS-8 range from 0-8, with scores of less than 6 reflecting low adherence.
Change from baseline to Month 12 in patient-reported Expanded Disability Status Scale (patient-reported EDSS) scores | Baseline and month 12
  The patient reported EDSS measures disability status on a scale ranging from 0 to 10, with higher scores indicating more disability. Scoring is based on measures of impairment in eight functional systems.
Proportion of patients relapsing at Month 12 | Month 12
  Relapses are defined as new or recurrent neurologic symptoms not associated with fever, lasting at least 24 hours.
Proportion of patients with relapses associated with hospitalizations at Month 12 | Month 12
Proportion of patients with relapses associated with steroid use at Month 12 | Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (10):
- Canada (10):
  - Research Site, Edmonton, Alberta
  - Research Site, Burnaby, British Columbia
  - Research Site, Saint John, New Brunswick
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Halifax, Nova Scotia
  - Research Site, Sydney, Nova Scotia
  - Research Site, Cambridge, Ontario
  - Research Site, London, Ontario
  - Research Site, Gatineau, Quebec
  - Research Site, Montreal, Quebec